CLINICAL TRIAL: NCT03078127
Title: Researching the Effects of Airway Clearance Therapies in Cystic Fibrosis (REACT-CF)
Brief Title: Researching the Effects of Airway Clearance Therapies in Cystic Fibrosis
Acronym: REACT-CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16-1813
Record Dates: First submitted 2017-02-27; First posted 2017-03-13 (Actual); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis; Mucociliary Clearance Defect
MeSH Terms: conditions — Cystic Fibrosis | interventions — BaseLine dental cement

STUDY DESIGN:
Intervention Model Description: All subjects will undergo baseline testing, followed by study procedures for three separate interventions, with subjects randomized into three arms in which a different sequence in which to complete the studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Sequence A (Active Comparator): In this arm, the interventions were performed in the following order:
  Baseline (prior to randomization), Whole body vibration, High Frequency Chest Wall Oscillation (HFCWO, aka "Vest" or TheVest®), Oscillatory Positive Expiratory Pressure (OPEP) (note this is different than the sequence shown in the example latin square shown in the included protocol, as that was meant to serve as an example -- actual randomization and formulation of the employed latin square / sequence generator was performed following completion of the protocol)
  Interventions: Other: Baseline (Huff-Cough alone); Device: Oscillatory Positive Expiatory Pressure Device; Device: Whole-Body Vibration Platform; Device: High Frequency Chest Wall Oscillatory Vest
- Sequence B (Active Comparator): In this arm, the interventions were performed in the following order:
  Baseline (prior to randomization), HFCWO, OPEP, Whole body vibration (note this is different than the sequence shown in the example latin square shown in the included protocol, as that was meant to serve as an example -- actual randomization and formulation of the employed latin square / sequence generator was performed following completion of the protocol)
  Interventions: Other: Baseline (Huff-Cough alone); Device: Oscillatory Positive Expiatory Pressure Device; Device: Whole-Body Vibration Platform; Device: High Frequency Chest Wall Oscillatory Vest
- Sequence C (Active Comparator): In this arm, the interventions were performed in the following order:
  Baseline (prior to randomization), OPEP, Whole body vibration, HFCWO (note this is different than the sequence shown in the example latin square shown in the included protocol, as that was meant to serve as an example -- actual randomization and formulation of the employed latin square / sequence generator was performed following completion of the protocol)
  Interventions: Other: Baseline (Huff-Cough alone); Device: Oscillatory Positive Expiatory Pressure Device; Device: Whole-Body Vibration Platform; Device: High Frequency Chest Wall Oscillatory Vest

INTERVENTIONS:
Other: Baseline (Huff-Cough alone) — Subjects will provide two "huffs" (forced expiratory maneuver with open glottis) followed by a cough every six minutes for a total of six Huff-Coughs.
Device: Oscillatory Positive Expiatory Pressure Device — Subjects will use an Areobika® branded OPEP device (10 breaths through highest tolerated resistance) prior to undergoing a Huff-Cough. Subjects will use the device six times every six minutes.
  Other Names: Aerobika
Device: Whole-Body Vibration Platform — Subjects will be seated on a PowerPlate® whole-body vibration platform for 90 seconds prior to Huff-Cough. Six intervals on the platform will be completed six minutes apart.
  Other Names: PowerPlate
Device: High Frequency Chest Wall Oscillatory Vest — Subjects will use TheVest® using a standardized "Minnesota Protocol" divided into six, four-minute segments, each followed by a Huff-Cough.
  Other Names: TheVest

SUMMARY:
This is a pilot study investigating the effectiveness and clinical efficacy of airway clearance therapy (ACT) in cystic fibrosis (CF). Enrolled subjects will undergo measurements of mucociliary clearance (MCC) and exhaled biomarkers at baseline and after 3 different forms of ACT: high frequency chest wall oscillatory vest, oscillatory positive expiratory pressure device, and whole-body vibration.

ELIGIBILITY:
Inclusion Criteria:

* Adults with confirmed diagnosis of cystic fibrosis aged 18 years and older.

Exclusion Criteria:

* Pregnant or lactating women,
* Individuals with severe lung disease (FEV1 <30%), or with exacerbations of lung disease requiring antibiotics or medication change within four weeks prior to enrolment.
* Individuals unable to use vest-based HFCWO, OPEP device, or who require oxygen supplementation at rest.
* Individuals with significant balance or gait impairment preventing them from tolerating being positioned on a vibrating platform.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron T Trimble, MD, Principal Investigator — Fellow; Scott Donaldson, MD, Principal Investigator — Associate Professor of Medicine
Locations (1):
- Marsico Clinical Research Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans at this time to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened and recruited from the adult CF clinic at UNC from January 2017 to December 2017.
Pre-assignment Details: Following screening, patients performed a baseline study visit prior to randomization into the study arms which determined which order to complete the other three interventions would be performed. Baseline (or "huff-cough") was completed prior to randomization to ensure comparator data if a patient was unable to complete the study.
Groups:
- Sequence A: In this arm, the interventions were performed in the following order:
  Baseline (prior to randomization), Whole body vibration, Vest, Oscillatory Positive Expiratory Pressure (OPEP).
  (note this is different than the sequence shown in the example latin square shown in the included protocol, as that was meant to serve as an example -- actual randomization and formulation of the employed latin square / sequence generator was performed following completion of the protocol)
- Sequence B: In this arm, the interventions were performed in the following order:
  Baseline (prior to randomization), Vest, OPEP, Whole body vibration (note this is different than the sequence shown in the example latin square shown in the included protocol, as that was meant to serve as an example -- actual randomization and formulation of the employed latin square / sequence generator was performed following completion of the protocol)
- Sequence C: In this arm, the interventions were performed in the following order:
  Baseline (prior to randomization), OPEP, Whole body vibration, Vest (note this is different than the sequence shown in the example latin square shown in the included protocol, as that was meant to serve as an example -- actual randomization and formulation of the employed latin square / sequence generator was performed following completion of the protocol)
Period: First Intervention
Arm/Group | Sequence A | Sequence B | Sequence C
Started | 4 | 3 | 3
Completed | 4 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Washout (3-21 Days)
Arm/Group | Sequence A | Sequence B | Sequence C
Started | 4 | 3 | 3
Completed | 4 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Sequence A | Sequence B | Sequence C
Started | 4 | 3 | 3
Completed | 4 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Washout (3-21 Days)
Arm/Group | Sequence A | Sequence B | Sequence C
Started | 4 | 3 | 3
Completed | 4 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Sequence A | Sequence B | Sequence C
Started | 4 | 3 | 3
Completed | 4 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adults with CF from the UNC adult CF center.
Groups:
- Sequence A: In this arm, the interventions were performed in the following order:
  Baseline (prior to randomization), Whole body vibration, Vest, OPEP (note this is different than the sequence shown in the example latin square shown in the included protocol, as that was meant to serve as an example -- actual randomization and formulation of the employed latin square / sequence generator was performed following completion of the protocol)
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Sequence C | Total
Number analyzed (Participants) | 4 | 3 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 3 | 10
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 42.25 [32 to 56] | 37.67 [21 to 57] | 41 [24 to 55] | 40.5 [21 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 3 | 3 | 2 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mucociliary Clearance-274
Description: As described in the protocol, gamma scintigraphy was used to measure clearance of particles from the whole right lung region of interest over 274 minutes. The primary outcome for this study was the area under the particle clearance curve from time 0 to 274 minutes post-inhalation (normalized to time by dividing by 274) and expressed as a percent, representing total average rate of mucociliary clearance (MCC).
Time Frame: 274 minutes
Measure: Mean (Standard Error); unit: percent clearance
Groups:
- Huff-Cough Alone: Subjects will provide two "huffs" (forced expiratory maneuver with open glottis) followed by a cough every six minutes for a total of six Huff-Coughs.
  Huff-Cough alone: Subjects will provide two "huffs" (forced expiratory maneuver with open glottis) followed by a cough every six minutes for a total of six Huff-Coughs.
- Oscillatory Positive Expiatory Pressure Device (OPEP): Subjects will use an Areobika® branded OPEP device (10 breaths through highest tolerated resistance) prior to undergoing a Huff-Cough. Subjects will use the device six times every six minutes.
  Oscillatory Positive Expiatory Pressure Device: Subjects will use an Areobika® branded OPEP device (10 breaths through highest tolerated resistance) prior to undergoing a Huff-Cough. Subjects will use the device six times every six minutes.
- Whole Body Vibration: Subjects will be seated on a PowerPlate® whole-body vibration platform for 90 seconds prior to Huff-Cough. Six intervals on the platform will be completed six minutes apart.
  Whole-Body Vibration Platform: Subjects will be seated on a PowerPlate® whole-body vibration platform for 90 seconds prior to Huff-Cough. Six intervals on the platform will be completed six minutes apart.
- High Frequency Chest Wall Oscillatory Vest (HFCWO): Subjects will use TheVest® using a standardized "Minnesota Protocol" divided into six, four-minute segments, each followed by a Huff-Cough.
  High Frequency Chest Wall Oscillatory Vest: Subjects will use TheVest® using a standardized "Minnesota Protocol" divided into six, four-minute segments, each followed by a Huff-Cough.
Arm/Group | Huff-Cough Alone | Oscillatory Positive Expiatory Pressure Device (OPEP) | Whole Body Vibration | High Frequency Chest Wall Oscillatory Vest (HFCWO)
Number analyzed (Participants) | 10 | 10 | 10 | 10
percent clearance | 20.3 (2.6) | 16.8 (3.1) | 18.5 (2.8) | 19.1 (2.3)
Statistical Analysis 1: Comparison: Huff-Cough Alone vs Oscillatory Positive Expiatory Pressure Device (OPEP) vs Whole Body Vibration vs High Frequency Chest Wall Oscillatory Vest (HFCWO); No comparable preliminary data exists on mucociliary clearance (MCC) in response to airway clearance therapy methods (ACTs) for a power calculation. However, prior studies of medication effect on MCC gave a baseline mean change of Ave270 clr of 27.7% (std dev of 15.1%). Thus, the investigators estimated a mean change of 20% for effective ACT with the same estimate for variability (Std Dev of 15.1%). Using a paired 2-tailed test to compare means, 7 subjects were estimated to be needed; Test type: Superiority; p = 0.615, ANOVA — ANOVA was performed (with multiple comparisons to compare each intervention to baseline) to assess for difference in MCC with each ACT. The a priori threshold for statistical significance was set to 0.05

2. Secondary Outcome: Mucociliary Clearance-90
Description: As described in the protocol, gamma scintigraphy was used to measure clearance of particles from the whole right lung region of interest over 274 minutes. This outcome for this study was the area under the particle clearance curve from time 0 to 90 minutes post-inhalation (normalized to time by dividing by 90) and expressed as a percent, representing average rate of mucociliary clearance (MCC) over 90 minutes.
Time Frame: 90 minutes
Population: All subjects were included for analysis
Measure: Mean (Standard Deviation); unit: percent clearance
Arm/Group | Huff-Cough Alone | Oscillatory Positive Expiatory Pressure Device (OPEP) | Whole Body Vibration | High Frequency Chest Wall Oscillatory Vest
Number analyzed (Participants) | 10 | 10 | 10 | 10
percent clearance | 13.8 (6.2) | 12.6 (5.9) | 12.4 (7.3) | 12.8 (6.9)
Statistical Analysis 1: Comparison: Huff-Cough Alone vs Oscillatory Positive Expiatory Pressure Device (OPEP) vs Whole Body Vibration vs High Frequency Chest Wall Oscillatory Vest; Test type: Superiority; p = 0.696, ANOVA — ANOVA was performed (with multiple comparisons to compare each intervention to baseline) to assess for difference in MCC with each ACT. The a priori threshold for significance was < 0.05

3. Secondary Outcome: Change in Rate of MCC
Description: Change in slope of particle clearance curve between pre intervention and ACT period.
Time Frame: pre-ACT (0-16 mins) and during ACT (16-50 mins)
Population: Only 4 subjects were included due to poor quality data obtained for slope measurement due to subject movement during the study (other MCC data used area under the curve data from key frames in which there was no subject movement, which proved to be more reliable). This data was not analyzed statistically.
Measure: Mean (Full Range); unit: %clearance / minute
Arm/Group | Huff-Cough Alone | Oscillatory Positive Expiatory Pressure Device (OPEP) | Whole Body Vibration | High Frequency Chest Wall Oscillatory Vest
Number analyzed (Participants) | 4 | 4 | 4 | 4
%clearance / minute | 0.011 [.001 to .023] | .013 [0.004 to 0.026] | 0.011 [-.004 to 0.027] | 0.010 [.001 to 0.017]

4. Secondary Outcome: Change in Fraction of Exhaled Nitric Oxide (FENO)
Description: FENO measurements were obtained pre- and post- intervention. The difference of post- vs pre- ACT FENO was reported.
Time Frame: pre and immediately post intervention (50 mins post inhalation)
Population: Only subjects who had measurable FENO above detection limits of the device (i.e. <5 ppm) for both before and after ACT were included in analysis. Data from subjects during interventions who did not have a detectable FENO for both pre- and post- ACT were excluded for analysis.
Measure: Mean (Standard Deviation); unit: ppm of NO
Arm/Group | Huff-Cough Alone | Oscillatory Positive Expiatory Pressure Device (OPEP) | Whole Body Vibration | High Frequency Chest Wall Oscillatory Vest
Number analyzed (Participants) | 8 | 8 | 6 | 6
ppm of NO | -1.84 (3.36) | -1.81 (2.65) | -1.42 (5.41) | -.75 (1.80)
Statistical Analysis 1: Comparison: Huff-Cough Alone vs Oscillatory Positive Expiatory Pressure Device (OPEP) vs Whole Body Vibration vs High Frequency Chest Wall Oscillatory Vest; The investigators compared FENO before and after ACT in a pooled manner (i.e., grouping each of the comparisons together), as the study was not powered for FENO comparisons within each ACT type; Test type: Superiority; p = 0.001, t-test, 2 sided — The a priori threshold of statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Huff-Cough Alone vs Oscillatory Positive Expiatory Pressure Device (OPEP) vs Whole Body Vibration vs High Frequency Chest Wall Oscillatory Vest; if the difference between pre and post-ACT FENO was significant (defined as p<0.05), it was investigated whether change in FENO correlated with MCC (as represented by Ave90Clr); Test type: Other — A linear regression was performed between change in FENO and Ave90Clr; p = 0.692, Regression, Linear — The a priori threshold for statistical significance (i.e., slope different than zero) between MCC and FENO was 0.05

5. Secondary Outcome: Purine Analysis (AMP) in Exhaled Breath Condensate
Description: Exhaled breath condensate was collected using a commercial device for this purpose. Concentrations of the purine adenosine monophosphate (AMP) and urea in this liquid were determined using mass spectrometry. This outcome was the difference in concentrations of AMP normalized to urea in this exhaled breath condensate between post-ACT and pre-ACT intervention.
Time Frame: pre and immediately post intervention (50 mins post inhalation)
Measure: Mean (Standard Deviation); unit: unitless ratio (AMP/Urea conc.)
Arm/Group | Huff-Cough Alone | Oscillatory Positive Expiatory Pressure Device (OPEP) | Whole Body Vibration | High Frequency Chest Wall Oscillatory Vest
Number analyzed (Participants) | 10 | 10 | 10 | 10
unitless ratio (AMP/Urea conc.) | -0.206 (0.679) | -.101 (0.124) | -.036 (0.650) | 0.144 (0.406)
Statistical Analysis 1: Comparison: Huff-Cough Alone vs Oscillatory Positive Expiatory Pressure Device (OPEP) vs Whole Body Vibration vs High Frequency Chest Wall Oscillatory Vest; The study was not designed or powered to assess for inter-group differences between the types of ACT, and for analytical purposes, these were pooled, with the analysis being a paired comparison within subjects to pre- to post-ACT; Test type: Superiority; p = 0.146, Wilcoxon signed-rank test — Non-parametric test used due to lack of data normality. The a prior threshold for statistical significance was < 0.05

6. Secondary Outcome: Purine Analysis (Adenosine) in Exhaled Breath Condensate (EBC)
Description: Difference of concentration of adenosine (a purine) in EBC between post-ACT and pre-ACT intervention.
Time Frame: pre and immediately post intervention (50 mins post inhalation)
Measure: Mean (Standard Deviation); unit: unitless ratio (adenosine/Urea conc.)
Arm/Group | Huff-Cough Alone | Oscillatory Positive Expiatory Pressure Device (OPEP) | Whole Body Vibration | High Frequency Chest Wall Oscillatory Vest
Number analyzed (Participants) | 10 | 10 | 10 | 10
unitless ratio (adenosine/Urea conc.) | -0.042 (0.166) | -0.027 (0.065) | -0.057 (0.134) | -.005 (0.057)
Statistical Analysis 1: Comparison: Huff-Cough Alone vs Oscillatory Positive Expiatory Pressure Device (OPEP) vs Whole Body Vibration vs High Frequency Chest Wall Oscillatory Vest; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.041, Wilcoxon signed-rank test — Non-parametric test used due to lack of data normality. The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Huff-Cough Alone vs Oscillatory Positive Expiatory Pressure Device (OPEP) vs Whole Body Vibration vs High Frequency Chest Wall Oscillatory Vest; If the difference between pre and post-ACT adenosine (purine) in EBC was significant (defined as p<0.05), the correlation between change in adenosine concentration and MCC (as represented by Ave90Clr) was investigated; Test type: Other — A linear regression was performed between change in pre and post-ACT adenosine (purine) in EBC and Ave90Clr; p = 0.047, Regression, Linear — The a priori threshold of statistical significance was p = 0.05

7. Secondary Outcome: Purine Analysis (Hypoxanthine) in Exhaled Breath Condensate
Description: Difference of concentration of hypoxanthine (a purine) in Exhaled Breath Condensate between post-ACT and pre-ACT intervention.
Time Frame: pre and immediately post intervention (50 mins post inhalation)
Measure: Mean (Standard Deviation); unit: unitless ratio (adenosine/Urea conc.)
Arm/Group | Huff-Cough Alone | Oscillatory Positive Expiatory Pressure Device (OPEP) | Whole Body Vibration | High Frequency Chest Wall Oscillatory Vest
Number analyzed (Participants) | 10 | 10 | 10 | 10
unitless ratio (adenosine/Urea conc.) | -1.04 (6.03) | -1.93 (4.16) | 1.64 (7.81) | 0.760 (1.88)
Statistical Analysis 1: Comparison: Huff-Cough Alone vs Oscillatory Positive Expiatory Pressure Device (OPEP) vs Whole Body Vibration vs High Frequency Chest Wall Oscillatory Vest; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.070, Wilcoxon signed-rank test — Non-parametric test used due to lack of data normality. The a priori threshold for statistical significance was < 0.05

ADVERSE EVENTS:
Time Frame: Screening for adverse event occurred from time of subject enrollment through completion and follow-up of all study procedures, up to a total of approximately 1 year.
Arm/Group | Huff-Cough Alone | Oscillatory Positive Expiatory Pressure Device (OPEP) | Whole Body Vibration | High Frequency Chest Wall Oscillatory Vest
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT03078127/Prot_SAP_000.pdf